CLINICAL TRIAL: NCT00625430
Title: A Phase I, Open-label, Dose Escalation Study to Assess the Safety and Tolerability of FP253 in Combination With Fludarabine Phosphate
Brief Title: A Phase I Gene Therapy Study of FP253/Fludarabine for Prostate Cancer
Acronym: FP253-GDEPT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotech Equity Partners Pty Ltd (Industry)
Responsible Party: Andrew M. Bray, Business Development Manager, Biotech Equity Partners Pty Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 253/001
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Gene Therapy; Fludarabine; Adenovirus; phase I
MeSH Terms: conditions — Prostatic Neoplasms; Adenoviridae Infections | interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Six Cohorts with escalating vector dose
  Interventions: Biological: Gene Directed Enzyme Prodrug Therapy, FP253/Fludarabine

INTERVENTIONS:
Biological: Gene Directed Enzyme Prodrug Therapy, FP253/Fludarabine — Subjects within a treatment group will be administered a single transrectal intraprostatic injection of FP253.
  Group A: 1 x 10Exp9 virus particles (VP); Group B: 3.2 x 10Exp9 VP; Group C: 1 x 10Exp10 VP; Group D: 3.2 x 10Exp10 VP; Group E: 1 x 10Exp11 VP; Group F: 3.2 x 10Exp 11 VP.
  If there are no dose-limiting toxicities, three additional patients may be treated at the highest dose.
  Twenty four hours following administration of the FP253, subjects will receive a first dose of fludarabine phosphate (20mg/m2 administered as an intravenous bolus). The first dose of fludarabine phosphate will be followed by 4 further doses at 24 hour intervals on treatment Days 3 to 6.
  Other Names: Fludarabine

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of a gene-directed enzyme prodrug therapy for prostate cancer. FP253 contains an ovine atadenovirus that expresses the E. coli enzyme purine nucleoside phosphorylase (PNP) under the control of a prostate-directed promoter. PNP converts systemically administered fludarabine (the prodrug) into 2-fluoroadenine (the active agent) at the site where FP253 has been administered (the prostate). This localized conversion is expected to provide organ-targeted chemotherapy that should reduce the systemic side effects associated with classical chemotherapy and also reduce the risk of debilitating damage to tissues surrounding the prostate.

DETAILED DESCRIPTION:
OBJECTIVES: The primary objective of this study is to determine the safety and tolerability of FP253 for prostate cancer. FP253 contains an ovine atadenovirus that expresses the E. coli enzyme purine nucleoside phosphorylase (PNP) under the control of a prostate-directed promoter.

SUBJECT POPULATION: Up to eighteen male subjects (6 groups of 3 subjects) who have a histological diagnosis of adenocarcinoma of the prostate, still have their prostate in situ, have evidence of progressive disease despite continuous androgen deprivation therapy and who meet all eligibility criteria, will be enrolled into this study.

STUDY DESIGN: This study is designed as an open-label, dose escalation trial in which each patient in a cohort will receive a single defined dose. Subjects will be enrolled consecutively into 6 escalating dose groups each of 3 subjects. Each subject will receive the treatment as outlined in the protocol and will be followed up for a further 2 years at regular intervals for life, as defined by current standard of care.

TREATMENT: Subjects will be administered a single injection of FP253 followed by five doses of Fludarabine phosphate as outlined in the Intervention section.

SAFETY PARAMETERS: Adverse events will be recorded and physical examinations, 12-lead ECG, vital sign monitoring, urinalysis and collection of blood samples for pathology laboratory tests will be performed at regular intervals during the study to monitor safety. The shedding of viral vector will be monitored as per regulatory requirement until negative.

ADDITIONAL PARAMETERS: In order to assess any haematological or immunological effects of this novel agent or any effects on tumour response and survival, the following will be assessed:

* Biochemical and Haematological Markers: including Prostate-Specific Antigen,
* Immunopathological Markers: including haematological markers and indicators of cytotoxicity,
* ECOG assessment,
* Assessment of disease progression and survival.

DATA ANALYSIS: Descriptive statistical methods will be used to summarize key data including demographics, vital sign measurements, ECG parameters, clinical laboratory parameters, immune response, tumour response, adverse events and concomitant medication. The general strategy of the safety analysis will be to examine the data summaries for any trends in safety parameters across the dose levels. No formal hypothesis will be tested.

A formal data analysis will be performed after all subjects have completed the study period (28 days) and an interim analysis will be performed after the first 3 dose cohorts have been completed. For the first year, three monthly follow up reports will be produced followed by 6 monthly reports for the second year and a final follow up report when all subjects have completed 2 years of follow up. Descriptive statistical methods will be used to summarise key data including demographics, vital sign measurements, ECG parameters, clinical laboratory parameters, immune response, tumour response, adverse events and concomitant medication. The general strategy of the safety analysis will be to examine the data summaries for any trends in safety parameters across the dose levels. No formal hypothesis will be tested.

ELIGIBILITY:
Inclusion Criteria (Prostate Cancer Categorization):

Subjects will have adenocarcinoma of the prostate which is progressive despite androgen deprivation therapy.

Subjects MUST fulfil each of the following criteria for inclusion in this study:

1. Biopsy of the tumour must have been performed and histological status of adenocarcinoma of the prostate documented. The diagnostic prostatic biopsy will have taken place at least 4 weeks prior to the planned day 1.
2. Subjects will have their prostate in situ.
3. Biochemical evidence of prostate cancer recurrence; defined as a rise over 3 successive PSA measurements spanning a minimum of 3 months (no lower limit of PSA exclusion).
4. Subjects will have been treated with androgen deprivation therapy and will remain on hormone therapy for the duration of the study (LHRH agonists with or without antiandrogens, or bilateral orchidectomy).
5. The Investigator should be able to localise the tumour either by digital rectal examination (DRE) (i.e. tumour palpable); or the tumour should be visible on transrectal ultrasound (TRUS). Localization of tumour will be documented and should be adequate to allow the Investigators to inject it. Repeated TRUS will be at the discretion of the Investigator General.

Inclusion Criteria (General):

Subjects MUST fulfil each of the following criteria for inclusion into this study:

1. Be male and be 18 years of age or greater.
2. Have voluntarily given written informed consent to participate in this study.
3. Have an ECOG performance status of 0, 1 or 2.
4. Have agreed to remain confined to the clinical testing facility for the first 3 days (2 nights) of the study.
5. Have adequate baseline organ function.
6. Have an ECG which is normal, or, if there is any abnormality, it must be considered to be clinically insignificant in the context of the trial.

Exclusion Criteria (Prostate Cancer Categorization):

Subjects with any of the following criteria will NOT be eligible for participation in this study:

1. Subjects who have had prior radical prostatectomy.
2. Subjects who are expected to die of prostate cancer within 3 months.

Exclusion Criteria (General):

Subjects with any of the following criteria will NOT be eligible for participation in this study:

1. Hypersensitivity to ciprofloxacin, fludarabine, pegfilgrastim or similar compounds.
2. Contraindications to fludarabine: subjects with decompensated haemolytic anaemia.
3. Contraindications to pegfilgrastim: known hypersensitivity to E. coli derived products.
4. Other associated or concomitant medical conditions that would interfere with the conduct of the study in the opinion of the treating physician.
5. Have used an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
6. Are immunocompromised or have used immunomodulatory agents/therapy within the 6 months preceding the initial treatment.
7. Subjects who, at the sole discretion of the Investigator, are judged to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events will be recorded. Physical examinations, 12-lead ECG, vital sign monitoring, urinalysis and collection of blood samples for pathology testing will be performed. Viral DNA and infectious virus will be monitored in serum and urine samples. | Selected assessments at Day: -14 (screening); Days: 1 to 6, 11, 15, 28; Months: 3, 6, 9, 12, 24

SECONDARY OUTCOMES:
Assess haematological and immunological markers, including Prostate-Specific Antigen (PSA) and C-ReactiveProtein (CRP). Effects on tumor response and survival. Immunopathological Markers. ECOG assessment. Assessment of disease progression and survival. | Selected assessments at Day: -14 (screening); Days: 1 to 6, 11, 15, 28; Months: 3, 6, 9, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: David N Dalley, MB BS FRACP, Principal Investigator — St Vincent's Hospital
Locations (1):
- St Vincent's Hospital, Sydney, Darlinghurst, New South Wales, Australia